CLINICAL TRIAL: NCT07046767
Title: A Multicenter Hybrid Platform Trial Comparing the Effects of a Prospective Cohort Treated With a Tri- Layer Amnion Graft or a Single Layer Amnion Graft to a Coarsened Exact Matched Retrospective Control Cohort of Patients With Hard-to-heal DFUs and VLUs
Brief Title: CAMP RWE Trial: Amnion Grafts for Healing Hard-to-Heal Ulcers in RW Populations
Acronym: CAMP RWE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capsicure, LLC (Network)
Collaborators: BioLab Holdings (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMP RWE
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Foot Ulcer (DFU); Venous Leg Ulcer; Wound; Foot
Keywords: DCF; VLU; Diabetic Foot Ulcer; Venus Leg Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Foot Injuries

STUDY DESIGN:
Intervention Model Description: This study will employ a platform umbrella design in which two studies will be run: one for diabetic foot ulcers and one for venous leg ulcers. Each study will have two intervention groups and one common SOC group.
  Subjects will be randomized to one of two interventions:
  IP1: BioLab Membrane Wrap Lite IP2: BioLab Tri-Membrane Wrap
  Subjects in the control group will be drawn from deidentified data sourced from the US Wound Registry. The US Wound Registry (USWR) is recognized by CMS as a Qualified Clinical Data Registry (QCDR). The matching of intervention to control groups will use coarsened exact matching (CSM) in which key variables are used to match: e.g., age, sex, baseline wound area, baseline wound age. The desired control subject pool should be three times larger than the prospective group (at least 165 in wound type).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): This study will employ a platform umbrella design in which two studies will be run: one for diabetic foot ulcers and one for venous leg ulcers. Each study will have two intervention groups and one common SOC group.
  Subjects will be randomized to one of two interventions:
  IP1: BioLab Membrane Wrap Lite IP2: BioLab Tri-Membrane Wrap
  Subjects in the control group will be drawn from deidentified data sourced from the US Wound Registry. The US Wound Registry (USWR) is recognized by CMS as a Qualified Clinical Data Registry (QCDR). The matching of intervention to control groups will use coarsened exact matching (CSM) in which key variables are used to match: e.g., age, sex, baseline wound area, baseline wound age. The desired control subject pool should be three times larger than the prospective group (at least 165 in wound type.)
- IP1: BioLab Membrane Wrap Lite (Experimental): This study will employ a platform umbrella design in which two studies will be run: one for diabetic foot ulcers and one for venous leg ulcers. Each study will have two intervention groups and one common SOC group.
  Subjects will be randomized to one of two interventions:
  IP1: BioLab Membrane Wrap Lite IP2: BioLab Tri-Membrane Wrap
  Subjects in the control group will be drawn from deidentified data sourced from the US Wound Registry. The US Wound Registry (USWR) is recognized by CMS as a Qualified Clinical Data Registry (QCDR). The matching of intervention to control groups will use coarsened exact matching (CSM) in which key variables are used to match: e.g., age, sex, baseline wound area, baseline wound age. The desired control subject pool should be three times larger than the prospective group (at least 165 in wound type.)
  Interventions: Other: IP1: BioLab Membrane Wrap Lite IP2: BioLab Tri-Membrane Wrap
- IP2: BioLab Tri-Membrane Wrap (Experimental): This study will employ a platform umbrella design in which two studies will be run: one for diabetic foot ulcers and one for venous leg ulcers. Each study will have two intervention groups and one common SOC group.
  Subjects will be randomized to one of two interventions:
  IP1: BioLab Membrane Wrap Lite IP2: BioLab Tri-Membrane Wrap
  Subjects in the control group will be drawn from deidentified data sourced from the US Wound Registry. The US Wound Registry (USWR) is recognized by CMS as a Qualified Clinical Data Registry (QCDR). The matching of intervention to control groups will use coarsened exact matching (CSM) in which key variables are used to match: e.g., age, sex, baseline wound area, baseline wound age. The desired control subject pool should be three times larger than the prospective group (at least 165 in wound type.)
  Interventions: Other: IP2: BioLab Tri-Membrane Wrap

INTERVENTIONS:
Other: IP1: BioLab Membrane Wrap Lite IP2: BioLab Tri-Membrane Wrap — BioLab Membrane Wrap LiteTM is a human tissue allograft derived from the amniotic membrane that provides structural tissue for use as a wound and protectant covering. Membrane Wrap LiteTM is a single-layer human tissue allograft, containing solely the amnion layer of Amniotic Membrane [Human Cellular and Tissue Based Product (HCT/P)] for transplantation regulated by the US Food and Drug Administration under 21 CFR Part 1271.
  Arms: IP1: BioLab Membrane Wrap Lite
Other: IP2: BioLab Tri-Membrane Wrap — BioLab Tri-Membrane WrapTM is a human tissue allograft derived from the amniotic membrane that provides structural tissue for use as a wound and protectant covering. Tri-Membrane WrapTM is a triple-layered human tissue allograft, containing amnion-chorion-amnion layers [Human Cellular and Tissue Based Product (HCT/P)] for transplantation regulated by the US Food and Drug Administration under 21 CFR Part 1271.
  Arms: IP2: BioLab Tri-Membrane Wrap

SUMMARY:
CAMP RWE Trial: A Multicenter hybrid platform trial comparing the effects of a prospective cohort treated with a tri-layer amnion graft or a single layer amnion graft to a coarsened exact matched retrospective control cohort of patients with hard-to-heal DFUs and VLUs

DETAILED DESCRIPTION:
A multicenter hybrid platform trial comparing the effects of a prospective cohort treated with a tri layer amnion graft or a single layer amnion graft to a coarsened exact matched retrospective control cohort of patients with hard-to-heal DFUs and VLUs

Hybrid prospective platform 2 arm, comparative, randomized multicenter study with a CSM matched retrospective control group Interventional comparative study

* IP 1: BioLab Membrane Wrap Lite
* IP2: BioLab Tri-Membrane Wrap

Standard of care: Debridement, maintenance of proper moisture balance, reduction in bacterial burden, offloading and multilayer compression.

Patients with nonhealing venous leg ulcerations or diabetic foot ulcers of at least 4-weeks duration that have failed to show 50% PAR with SOC therapies Patients receiving SOC therapies for hard-to-heal VLUs and/or DFUs

To gather prospective real-world evidence (RWE) in both diabetic foot ulcers and venous leg ulcers increasing the understanding of treatment performance in everyday clinical settings, capturing insights from a more diverse patient population than traditional clinical trials. This information is vital for evaluating the effectiveness of innovative wound care strategies in practical, real-life scenarios

To demonstrate the clinical effectiveness of IP1 and IP2 as an adjunct to standard of care in supporting wound healing compared to standard of care alone in venous leg ulcers and diabetic foot ulcers across the continuum of care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age and older
2. 2. Subjects having a non-healing venous leg ulcer or diabetic foot ulcer of >4 weeks duration and visible signs of healing objectively, less than 50% reduction in wound size in the last 4 weeks
3. Subjects' wound size is minimum of 2 cm2 and maximum of 25cm2
4. If the subject has more than one eligible wound the largest wound will be selected (the index wound)
5. Subject is able and willing to follow the protocol requirements
6. Subject has signed informed consent

Exclusion Criteria:

1. Inability to adhere to the study protocol or study visit schedule
2. Pregnancy
3. Child-bearing potential without appropriate contraception
4. Lactation
5. Treatment of the wound with engineered tissue or other scaffold materials within 30 days preceding the first treatment visit.
6. Visible signs of improvement in the four weeks before randomisation (defined objectively as a 50% reduction in surface area in the four weeks before enrolment)
7. The subject has other concurrent conditions that in the opinion of the investigator may compromise subject safety
8. Known contraindications to the use of amniotic tissue grafts
9. The index ulcer shows clinical signs and symptoms of wound infection needing treatment with local or systemic antimicrobials or antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Wound Closure | 12 Weeks
  To demonstrate the clinical effectiveness of IP1 and IP2 as an adjunct to standard of care in supporting wound healing compared to standard of care alone in venous leg ulcers and diabetic foot ulcers across the continuum of care. Thus, the incidence of index ulcers obtaining complete wound closure by 12 weeks will be collected.

SECONDARY OUTCOMES:
Wound percent area reduction | Weeks 4, 8, and 12
  To demonstrate real world utilization and utility of two novel amniotic tissue grafts to support a variety of meaningful clinical outcomes in an at-risk patient population this study will collect wound percent area reduction at 4, 8, 12 weeks, change from baseline in quality of life, based on changes in index wound quality of life Wound-Q, and subject pain scores.

CONTACTS AND LOCATIONS:
Overall Officials: Windy Cole, DPM, Study Director — Capsicure, LLC
Locations (7):
- United States (7):
  - FOMAT Medical Research, Oxnard, California
  - Solutions Medical Research, Coral Gables, Florida
  - Nova Medical Services - Research Division LLC, Miami, Florida
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - St. Louis Foot and Ankle, LLC, St Louis, Missouri
  - Jevlos Health, Inc, Syosset, New York
  - Hope Vascular and Podiatry, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the study sponsor. Any investigator involved with this study is obligated to provide the sponsor with complete test results and all data derived from the study.